CLINICAL TRIAL: NCT02276027
Title: A Phase II, Open Label, Multiple Arm Study of Single Agent AUY922, BYL719, INC280, LDK378 and MEK162 in Chinese Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase II, Open Label, Multiple Arm Study of AUY922, BYL719, INC280, LDK378 and MEK162 in Chinese Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2205
Record Dates: First submitted 2014-10-09; First posted 2014-10-27 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Adenocarcinoma Lung Cancer; Squamous Cell Lung Carcinoma
Keywords: adenocarcinoma lung cancer,; squamous cell lung carcinoma,; NSCLC
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Alpelisib; capmatinib; ceritinib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BYL719 350 mg QD (Experimental): Patient's tumor must have molecular alteration of the PIK3CA gene.
  Interventions: Drug: BYL719
- INC280 400 mg BID tab/600 mg BID cap (Experimental): Patient's tumor must have molecular alteration of the c-MET gene.
  Interventions: Drug: INC280
- LDK378 750 mg QD (Experimental): Patient's tumor must have ALK or ROS1 gene rearrangement.
  Interventions: Drug: LDK378
- MEK162 45 mg BID (Experimental): Patient's tumor must have KRAS, NRAS or BRAF mutation.
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: BYL719 — BYL719 was dosed as 350 mg once daily. On the first day of each cycle, patient received a prescription of adequate drug supply for self-administration at home. The investigator must emphasized compliance and instructed the patient to take BYL719 exactly as prescribed.
  Arms: BYL719 350 mg QD
Drug: INC280 — INC280 was dosed as 600 mg (tablet) or 400mg(Capsule) twice daily. On the first day of each cycle, patient received a prescription of adequate drug supply for self-administration at home. The investigator must emphasized compliance and instructed the patient to takeINC280 exactly as prescribed.
  Arms: INC280 400 mg BID tab/600 mg BID cap
Drug: LDK378 — LDK378 was dosed as 750 mg once daily. On the first day of each cycle, patient received a prescription of adequate drug supply for self-administration at home. The investigator must emphasized compliance and instructed the patient to take LDK378 exactly as prescribed.
  Arms: LDK378 750 mg QD
Drug: MEK162 — MEK162 was dosed as 45 mg twice daily. On the first day of each cycle, patient received a prescription of adequate drug supply for self-administration at home. The investigator must emphasized compliance and instructed the patient to take MEK162 exactly as prescribed.
  Arms: MEK162 45 mg BID

SUMMARY:
The purpose of this study was to evaluate the anti-tumor activity of single agent BYL719, INC280, LDK378 and MEK162 in advanced NSCLC patients carrying specific molecular alterations.

There is a great unmet medical need in NSCLC patients with advanced or metastatic disease. Novel approaches using targeted therapeutic agents for these patient populations with molecular characterization could potentially identify subsets of advanced NSCLC patients who would benefit from targeted kinase inhibition. Study treatments, BYL719, INC280, LDK378 and MEK162, which target PIK3CA, c-MET, ALK/ROS1 and MEK respectively, have shown promising data in either preclinical or clinical lung cancer settings.

DETAILED DESCRIPTION:
To enter the screening phase of the study, the subjects' molecular alterations were determined using locally validated methodologies from a newly obtained tumor sample (preferred) or the most recent archival tumor sample available. Based on the molecular alterations of the tumor, subjects were assigned to one of the treatment arms. Subjects with multiple molecular alterations in epidermal growth factor receptor (EGFR) and the relevant pathways were excluded, except under the conditions described in Inclusion criteria.

The treatment period began on Cycle 1 Day 1 and continued in 28-day cycles until disease progression, unacceptable toxicity, withdrawal of informed consent, death or the subject transferred to another Novartis study that could continue to provide the study drug.

All subjects were required to be followed up for 30 days for safety after receiving the last dose of study treatment. Subjects who discontinued study treatment for any reason other than disease progression were followed up for progression of disease. All subjects were required to be followed for survival. For subjects transferred to another Novartis study, an end of treatment visit (EOT) was required to be performed and the subject would not enter the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (stage IIIB or stage IV) NSCLC
* Must have specific molecular alterations

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases which are neurologically unstable or requiring increasing doses of steroids within the 4 weeks prior to study entry to control their CNS disease
* Radiation therapy within ≤ 4 weeks prior to study entry, with the exception of limited field palliative radiotherapy for bone pain relief.
* Any other malignancies within the last 5 years before study entry
* Major surgery ≤ 2 weeks prior to study entry or who have not recovered from side effects of such therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from China
Pre-assignment Details: To enter the screening phase, the subjects' molecular alterations were determined using locally validated methodologies from a newly obtained tumor sample or the most recent archival tumor sample available. Based on the molecular alterations of the tumor, subjects were assigned to one of the treatment arms. Subjects with multiple molecular alterations in epidermal growth factor receptor and the relevant pathways were excluded, except under the conditions described in Inclusion criteria.
Period: Overall Study
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Started | 2 | 16 | 26 | 22
Completed | 0 | 0 | 6 | 0
Not Completed | 2 | 16 | 20 | 22
Not completed — Death | 1 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Progressive disease | 1 | 13 | 12 | 14
Not completed — Subject/guardian decision | 0 | 1 | 0 | 3
Not completed — Adverse Event | 0 | 2 | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID | Total
Number analyzed (Participants) | 2 | 16 | 26 | 22 | 66
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 53.0 [44 to 62] | 58.2 [47 to 65] | 49.4 [33 to 66] | 60.3 [48 to 74] | 55.3 [33 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 15 | 3 | 23
  Male | 2 | 11 | 11 | 19 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is the proportion of patients with a best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria (Overall Response (OR) = CR + PR).
  Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 231 weeks
Population: Full analysis set: all subjects who received at least one dose of the respective study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 16 | 26 | 22
Participants | 0 | 3 | 19 | 2

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS is defined as the time from date of randomization/start of treatment to date of death due to any cause.
Time Frame: Up to 231 weeks
Population: Full analysis set: all subjects who received at least one dose of the respective study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 16 | 26 | 22
Months | 4.99 [0.30 to 9.69] | 13.26 [1.18 to 23.33] | NA [19.35 to NA] — Median and upper limit NA because they are not evaluable. The median OS was not reached | 9.20 [3.52 to 11.93]

3. Secondary Outcome: Number of Participants With Progression-free Survival (PFS)
Description: PFS event is defined as the first documented progression or death due to any cause according to RECIST 1.1 criteria
Time Frame: Up to 231 weeks
Population: Full analysis set: all subjects who received at least one dose of the respective study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 16 | 26 | 22
Participants | 2 | 16 | 19 | 19

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is the percentage of patients with a best overall response of complete response (CR) or partial response (PR) or Stable Disease (SD) according to RECIST 1.1 criteria (DCR: CR+PR+SD) Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD
Time Frame: Up to 231 weeks
Population: Full analysis set: all subjects who received at least one dose of the respective study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 16 | 26 | 22
Percentage of participants | 50.0 [1.3 to 98.7] | 43.8 [19.8 to 70.1] | 92.3 [74.9 to 99.1] | 59.1 [36.4 to 79.3]

5. Secondary Outcome: Median Duration of Overall Response (DOR)
Description: Duration of overall response (DOR) is defined as the time from the first documented CR or PR (confirmed by the subsequent assessment) to the date of the first documented progression or death due to underlying cancer.
Time Frame: Up to 231 weeks
Population: Full analysis set subjects with confirmed complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 0 | 3 | 19 | 2
Months |  | 3.84 [3.81 to 5.59] | 34.96 [7.59 to NA] — Upper limit NA because it is not evaluable | 5.47 [3.55 to 7.39]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
  If CTCAE grading does not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, corresponding to grades 1 - 4, was used.
Time Frame: up to 235 weeks
Population: Safety Set: Includes all patients who received at least one dose of the respective study medication and had at least one valid postbaseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 16 | 26 | 22
Participants
  AE All grades | 2 | 16 | 26 | 22
  AE Grade 3/4 | 1 | 11 | 23 | 20
  SAE All grades | 1 | 12 | 11 | 18
  SAE Grade 3/4 | 1 | 7 | 9 | 15

7. Secondary Outcome: Pharmacokinetics Profile, AUCtau and AUClast
Description: PK parameters are estimated from each individual plasma concentration-time profile using non-compartmental analysis (Phoenix software version 6.2 and above).
  AUCtau is the AUC calculated to the end of a dosing interval (tau) (amount x time x volume-1) AUClast is the AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1) On Cycle 1 Day 1, PK parameters for only BYL719 350 mg QD arm were analyzed
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours) and Day 15 (pre dose, 0.5, 1, 2, 4, 6, 8 hours post dose and only for BYL719 350 mg QD and LDK378 750 mg QD arms also at 24 hours post dose)
Population: PAS: Pharmacokinetic analysis set includes all subjects who have at least one blood sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 14 | 6 | 9
ng*h/mL
  AUClast Cycle 1 Day 1: number analyzed (Participants) | 2 | 0 | 0 | 0
  AUClast Cycle 1 Day 1 | 20909 (107) |  |  |
  AUCtau Cycle 1 Day 15: number analyzed (Participants) | 1 | 14 | 6 | 9
  AUCtau Cycle 1 Day 15 | 23892 (NA) — SD is NA since there is only 1 subject with evaluable PK profile | 32034 (6992) | 30361 (3807) | 2645 (981)
  AUClast Cycle 1 Day 15: number analyzed (Participants) | 1 | 14 | 6 | 9
  AUClast Cycle 1 Day 15 | 23721 (NA) — SD is NA since there is only 1 subject with evaluable PK profile | 27875 (7629) | 28013 (5006) | 2642 (1026)

8. Secondary Outcome: Pharmacokinetics Profile, Cmax
Description: PK parameters are estimated from each individual plasma concentration-time profile using non-compartmental analysis (Phoenix software version 6.2 and above).
  Cmax is the maximum (peak) observed plasma concentration (mass x volume-1) On Cycle 1 Day 1, PK parameters for only BYL719 350 mg QD arm were analyzed
Time Frame: as for outcome 7
Population: PAS: Pharmacokinetic analysis set includes all subjects who have at least one blood sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 14 | 6 | 9
ng/mL
  Cmax Cycle 1 Day 1: number analyzed (Participants) | 2 | 0 | 0 | 0
  Cmax Cycle 1 Day 1 | 2135 (700) |  |  |
  Cmax Cycle 1 Day 15: number analyzed (Participants) | 1 | 14 | 6 | 9
  Cmax Cycle 1 Day 15 | 2630 (NA) — SD is NA since there is only 1 subject with evaluable PK profile | 8046 (3550) | 1362 (177) | 587 (183)

9. Secondary Outcome: Pharmacokinetics Profile, Tmax
Description: PK parameters are estimated from each individual plasma concentration-time profile using non-compartmental analysis (Phoenix software version 6.2 and above).
  Tmax is the time to reach maximum (peak) plasma concentration (time) On Cycle 1 Day 1, PK parameters for only BYL719 350 mg QD arm were analyzed
Time Frame: as for outcome 7
Population: PAS: Pharmacokinetic analysis set includes all subjects who have at least one blood sample providing evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
Number analyzed (Participants) | 2 | 14 | 6 | 9
hours
  Tmax Cycle 1 Day 1: number analyzed (Participants) | 2 | 0 | 0 | 0
  Tmax Cycle 1 Day 1 | 4.03 [2.05 to 6.00] |  |  |
  Tmax Cycle 1 Day 15: number analyzed (Participants) | 1 | 14 | 6 | 9
  Tmax Cycle 1 Day 15 | 2.00 [2.00 to 2.00] | 1.00 [0.467 to 6.17] | 6.10 [2.03 to 8.00] | 1.10 [0.517 to 7.58]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days after receiving the last dose of study treatment, up to maximum duration of 235 weeks.
Description: Any sign or symptom that occurs during the study treatment plus 30 days after receiving the last dose of study treatment.
Arm/Group | BYL719 350 mg QD | INC280 400 mg BID Tab/600 mg BID Cap | LDK378 750 mg QD | MEK162 45 mg BID
All-Cause Mortality (participants affected / at risk) | 1/2 | 4/16 | 1/26 | 5/22
Serious Adverse Events (participants affected / at risk) | 1/2 | 12/16 | 11/26 | 18/22
Other Adverse Events (participants affected / at risk) | 2/2 | 16/16 | 26/26 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYL719 350 mg QD (N=2) | INC280 400 mg BID Tab/600 mg BID Cap (N=16) | LDK378 750 mg QD (N=26) | MEK162 45 mg BID (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Rheumatic heart disease (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 4
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYL719 350 mg QD (N=2) | INC280 400 mg BID Tab/600 mg BID Cap (N=16) | LDK378 750 mg QD (N=26) | MEK162 45 mg BID (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 13 | 19 | 18
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular dissociation (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 5 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Wandering pacemaker (Cardiac disorders) | 0 | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 7 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 2 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 3 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 11 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 20 | 3
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 26 | 14
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3 | 5
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 2 | 8
Nausea (Gastrointestinal disorders) | 0 | 6 | 12 | 6
Oesophageal oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 6 | 20 | 9
Asthenia (General disorders) | 0 | 2 | 10 | 7
Chest discomfort (General disorders) | 1 | 5 | 5 | 2
Chills (General disorders) | 0 | 1 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 5
Fatigue (General disorders) | 0 | 2 | 3 | 3
Impaired healing (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 5 | 12 | 2
Oedema peripheral (General disorders) | 0 | 5 | 4 | 11
Pain (General disorders) | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 5 | 7 | 10
Sensation of foreign body (General disorders) | 0 | 1 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Erythrasma (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 3 | 2 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 5 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 7 | 24 | 6
Albumin urine present (Investigations) | 0 | 3 | 0 | 0
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2
Amylase increased (Investigations) | 0 | 7 | 8 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 5 | 26 | 16
Bilirubin conjugated increased (Investigations) | 0 | 3 | 7 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 5 | 15 | 6
Blood bilirubin increased (Investigations) | 0 | 5 | 3 | 3
Blood cholesterol increased (Investigations) | 1 | 2 | 2 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 7 | 16
Blood creatinine increased (Investigations) | 1 | 7 | 10 | 0
Blood fibrinogen increased (Investigations) | 0 | 2 | 0 | 0
Blood glucose increased (Investigations) | 0 | 2 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 2 | 4 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 2 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 10 | 6
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 1 | 0
Enzyme level increased (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 9 | 15 | 4
Glucose urine present (Investigations) | 0 | 2 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 0 | 2 | 5 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0
PO2 decreased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 1 | 1 | 3
Protein urine present (Investigations) | 0 | 1 | 2 | 2
Prothrombin time prolonged (Investigations) | 0 | 1 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Thrombin time prolonged (Investigations) | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 0 | 1 | 15 | 1
Weight increased (Investigations) | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 2 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9 | 14 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5 | 9 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 7 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5 | 17 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 14 | 21 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 4 | 8
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 8 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 6 | 9 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 8 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 5 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 12 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 9 | 4
Dreamy state (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 6 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 3 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 4 | 2
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0
Tic (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 17 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 6 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 9 | 3
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 12 | 16
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 4
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT02276027/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT02276027/SAP_001.pdf